CLINICAL TRIAL: NCT06230536
Title: Contribution of High-resolution Manometry With Impedancemetry for the Evaluation of Esophageal Clearance in Achalasia
Brief Title: MARIMPACH : Contribution of High-resolution Manometry With Impedancemetry for the Evaluation of Esophageal Clearance in Achalasia
Acronym: MARIMPACH
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2023/55
Record Dates: First submitted 2024-01-19; First posted 2024-01-30 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Esophageal Achalasia
Keywords: timed baryum esophagogram; high-resolution manometry with impedancemetry; esophageal clearance; Eckardt score
MeSH Terms: conditions — Esophageal Achalasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Outcome after treatment of achalasia is usually assessed by the Eckardt score (ES). The timed barium esophagogram (TBE) is used to objectively assess esophageal clearance after treatment. High-resolution manometry with impedancemetry (HRiM) provides information on esophageal clearance of liquids in addition to motility parameters. The aim of this study was to compare esophageal clearance determined by HRiM and TBE in patients with achalasia treated by POEM.

DETAILED DESCRIPTION:
Consecutive patients treated with POEM had pre and post-POEM assessment with ES, TBE, and HRiM. Treatment failure was defined by an ES > 3 at 3 months post-POEM. Incomplete esophageal clearance (IEC) was defined by the presence of an esophageal stasis > 2 cm at 5 minutes in HRiM and/or TBE. The Eckardt score is evaluated at one year to estimate the prognostic value of measurements of esophageal clearance after treatment on long-term symptoms. The evaluation of the Eckardt score will be compared to the quality of life score. All of these examinations are carried out as part of routine care.

The supposed superiority of HRiM in the evaluation of esophageal clearance, systematically carried out in the assessment of Achalasia, could lead to no longer using TBE which is a irradiating examination for the patient.

ELIGIBILITY:
Inclusion Criteria:

* The patients included are all patients treated by POEM at Bordeaux University Hospital between October 2020 and September 2024.

Exclusion Criteria:

* Primary POEM failure, lost to follow-up, absence of completion of the ES, TBE or HRiM pre or post poem at 3 months.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: a single cohort of all patients with achalasia and treated by POEM at Bordeaux University Hospital and having performed HRiM and TBE in routine care
Sampling Method: Non-Probability Sample
Enrollment: 104 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
esophageal clearance | 3 months
  Difference of esophageal clearance determined by HRiM and TBE in patients with achalasia treated by POEM at 3 months

SECONDARY OUTCOMES:
Efficacy : score of Eckardt | 3 months, 12 months
  Evaluation of Eckardt score at 3 months and 12 months post-POEM . Each question is rated from 0 to 3. It consists of 4 items with a total score varies from 0 to 12.
Efficacy : esophageal clearance | 3 months
  Evaluation of esophageal clearance at 3 months post-POEM .
Quality of life : Score QLQ-SF36 | 3 months
  Self-questionnaire in 36 items evaluating the quality of life. The SF-36 questionnaire is made up of 36 questions which concern the last four weeks, divided into 8 dimensions (Physical activity / Life and relationships with others / Physical pain / Perceived health / Vitality / Limitations due to psychological state / Limitations due to physical state / Mental health).
Quality of life : QLQ-OES24 | 3 months
  The QLQ-OES24 consists of 24 items assessing dysphagia, deglutition, abdominal/GI symptoms, eating difficulties, pain, emotional problems relating to esophageal cancer and to side effects of chemotherapy/radiotherapy.
Quality of life : GERD-HRQL | 3 months
  The GERD-HRQL was developed to survey symptomatic outcomes and therapeutic effects in patients with GERD. The scale has 11 items, which focus on heartburn symptoms, dysphagia, medication effects and the patient's present health condition.
Quality of life : ASQ (Achalasia Quality of Life) | 3 months
  The ASQ is a validated 10 questions questionnaire where patients can quantify and qualify symptoms of achalasia such as dysphagia to both solids and liquids, specific types of food, other associated symptoms, and overall health in relation to achalasia.
Quality of life : RDQ (Reflux Disease Questionnaire): | 3 months
  The RDQ is a questionnaire in which subjects are asked to report the frequency and severity of their upper gastrointestinal symptoms (six items). There are three subscales that evaluate regurgitation, heartburn, and dyspepsia. The heartburn and regurgitation subscales can be combined into a GERD dimension.

CONTACTS AND LOCATIONS:
Overall Officials: Arthur BERGER, MD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Chu de Bordeaux, Pessac, France

IPD SHARING:
Plan to Share IPD: No